CLINICAL TRIAL: NCT04969718
Title: Suicide Prevention by Empowering Adolescents in Pakistan (SEPAK): A Feasibility Study for Research Capability and Trial Readiness in Pakistan
Brief Title: Suicide Prevention by Empowering Adolescents in Pakistan (SEPAK)
Acronym: SEPAK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pakistan Institute of Living and Learning (Other)
Collaborators: University of Manchester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: SEPAK
Record Dates: First submitted 2021-07-05; First posted 2021-07-21 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Self-harm
Keywords: self-harm; suicide prevention; school-based intervention; Pakistan
MeSH Terms: conditions — Self-Injurious Behavior; Suicide Prevention | interventions — Lead; Referral and Consultation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- LEADS Plus educational posters (Experimental): A total of six group sessions with students using presentations and videos.
  Interventions: Other: LEADS Plus educational posters; Other: educational posters
- Question, Persuade, and Refer (Teachers) Plus educational posters (Experimental): It is a manualised programme for gatekeepers (teachers). This includes both presentations and videos.
  Interventions: Other: Question, Persuade, and Refer (Teachers) Plus educational posters; Other: educational posters
- Screening by Professionals programme Plus educational posters (Experimental): This is an indicated or selective intervention by health professionals who will review assessments (done using structured questionnaires) and refer students where necessary.
  Interventions: Other: Screening by Professionals programme plus educational posters; Other: educational posters
- Educational poster (Active Comparator): The control group will be exposed to the six educational posters.
  Interventions: Other: educational posters
- Question, Persuade, and Refer (Parents) Plus educational posters (Experimental): It is a manualised programme for gatekeepers (parents). This includes both presentations and videos.
  Interventions: Other: educational posters; Other: Question, Persuade, and Refer (Parents) Plus educational posters

INTERVENTIONS:
Other: LEADS Plus educational posters — This intervention covers depression and its symptoms, the link between depression and suicide, the risk and protective factors associated with suicide, the warning signs of suicide, seeking help and overcoming barriers to seeking help, and school and community suicide prevention resources. Six educational posters will also be displayed in class rooms
  Arms: LEADS Plus educational posters
Other: Question, Persuade, and Refer (Teachers) Plus educational posters — It is a manualised programme for gatekeepers, originally developed in the USA which to train teachers/school staff to identify the suicide risk in students and encourage students at risk of suicide to seek professional help. Six educational posters will also be displayed in classrooms.
  Arms: Question, Persuade, and Refer (Teachers) Plus educational posters
Other: Screening by Professionals programme plus educational posters — This is an indicated or selective intervention which is based on students' responses to the baseline questionnaires. Participating health professionals review students' responses to the questionnaires used in the study and students whose scores meet pre-established cutoff points will be invited to participate in a professional mental health clinical assessment and if needed, referred to clinical services. Six educational posters will also be displayed in classrooms.
  Arms: Screening by Professionals programme Plus educational posters
Other: educational posters — Six educational posters will be displayed in all schools in this cluster.
Other: Question, Persuade, and Refer (Parents) Plus educational posters — It is a manualised programme for gatekeepers (parents), originally developed in the USA which to train parents to support the young people at risk of suicide. Six educational posters will also be displayed in classrooms.
  Arms: Question, Persuade, and Refer (Parents) Plus educational posters

SUMMARY:
Self-harm is now seen as an epidemic affecting young people across the world and particularly in low and middle-income countries (LMIC) such as Pakistan. Young people in Pakistan often come across many troubles such as mental health and family problems, stress at school and social and economic inequalities. A youth suicide prevention programme is needed in Pakistan. Such programme will be based on secondary schools (where most young people are) and will support schools to work together with many public agencies to tackle the full range of troubles that young people face. Our main research aim is to work together with multiple stakeholders to culturally adapt and test the feasibility of three SEPAK interventions to prevent suicide among students in secondary schools in Pakistan (aged 12 to 17 years).

DETAILED DESCRIPTION:
There will be two research phases. In the first phase,

1. Four preventative interventions will be selected and translated after reviewing the international literature on youth suicide prevention programmes (e.g. SEYLE trial in Europe);
2. Focus groups will be undertaken with multiple stakeholders (students, teachers/staff at secondary schools, parents and health professionals) to decide on adaptations needed to the four selected interventions;
3. Adapted versions the four preventative SEPAK interventions will be produced after incorporating the modifications recommended by the focus groups with stakeholders.

In the second phase, the feasibility and acceptability of the four preventative SEPAK interventions will be examined in 4 secondary schools (each site) and one control group (each site) across 8 cities in Pakistan. The four preventative interventions will involve i. Delivering workshops for students at secondary schools to raise awareness on mental health and stresses that students face.

ii. Training school teachers/workers to act as facilitators and identify troubled students iii. Training parents to act as facilitators and identify and support troubled young people iv. Training of health professionals who work with young people to systematically use cut-off scores of established psychometric tools for referring young people to mental and social care services. Six posters on mental health awareness will display in the classrooms of the school allocated to the control group.

ELIGIBILITY:
Inclusion Criteria for students:

1. age 12 - 17 years
2. the school authority agrees for the student to participate;
3. both parents and students willing to participate.

Exclusion Criteria students:

1. the school authority refuses for the student to participate;
2. the adolescents attend a specialist and/or independent or private school;
3. the parents of students in a participating school, or the students themselves, have refused to sign the consent document.

Parents/guardians

Parents/guardians are eligible to participate if they meet all the following criteria:

1. caring for pupils aged 12-17 years;
2. the school authority agrees for the school to participate;
3. willing to participate in the study;
4. willing for pupils they care for to participate in the baseline and post-intervention assessments.

If parents/guardians meet the following exclusion criteria, they are ineligible to participate:

1. the school authority refuses for the school to participate;
2. the pupils they care for attend a specialist and/or independent or private school;
3. not willing to participate in the study or not willing for the pupils they care for to participate in the baseline and post-intervention assessments.

Inclusion criteria (schools)

1. the school authority agrees to participate;
2. the schools shall be non-specialist public schools;
3. school contains at least 80 students;
4. school has more than 3 teachers;
5. no more than 60% of students are of either sex;
6. informed consent from parents and students is obtained.

Exclusion criteria (schools)

1. the school authority refuses to participate;
2. the adolescents attend a specialist and/or independent or private school;

Inclusion criteria (Health Professionals)

Health professionals are eligible to participate if they meet all the following criteria:

1. Health professionals practicing within selected union councils
2. Willing to participate in the study Exclusion criteria (health professionals)

(1) Health professionals not currently practicing within selected union councils (2) Not willing to participate in the study

Teachers/staff at schools

Teachers and other school staff are eligible to participate if they meet all the following criteria:

1. working with pupils aged 12-17 years;
2. their school authority agrees for the school to participate;
3. willing to participate in the study;

If teachers and staff at school meet the following exclusion criteria; they are ineligible to participate:

1. their school authority refuses for the school to participate;
2. not willing to participate in the study

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1350 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-04-28 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Feasibility of undertaking a trial of the intervention | Change from baseline to 1-month post baseline
  recruitment rate of the trial
Therapy log | Change from baseline to 1-month post baseline
  acceptability of the interventions that will be evident from the attendance of participants in each session on a therapy log

SECONDARY OUTCOMES:
The Global school-based student health survey (GSHS) | Change in scores from baseline to outcome (1-month post baseline)
  The is a self-administered questionnaire and covered ten key topics: alcohol use, dietary behaviors, drug use, hygiene, mental health, physical activity, protective factors, sexual behaviors, tobacco use, and violence and unintentional injury
Deliberate Self-Harm Inventory | Change in scores from baseline to outcome (1-month post baseline)
  DSHI will be used to collect information about episode of self-harm. Minimum score is 0 and maximum score is 34. Higher total score indicate the higher intensity of the problem.
Kessler Psychological Distress Scale | Change in scores from baseline to outcome (1-month post baseline)
  This will use to measure psychological distress. It's a 10 item scale measuring emotional states with a 5 level response scale. Minimum score is 10 and a maximum score is 50. Low scores indicate low levels of psychological distress and high scores indicate high levels of psychological distress.
Beck Scale for Suicidal Ideation (BSSI) | Change in scores from baseline to outcome (1-month post baseline)
  This scale is a 19-items instrument that evaluates the presence and intensity of suicidal thoughts in a week. Minimum total score is 0 and maximum total score can be 38. Higher scores indicate worse outcome.
Euro-Qol (EQ-5D-5L) | Change in scores from baseline to outcome (1-month post baseline)
  A standardised instrument to measure health status and associated population utility weights. It consists of a self-report questionnaire covering five dimensions of health (mobility, self-care, usual activities, pain/ discomfort and anxiety/ depression)
Client Service Receipt Inventory | Change in scores from baseline to outcome (1-month post baseline)
  We will collect information on the use of health services (including the informal sector such as faith healers/Imams)
Client Satisfaction Questionnaire | Scores reported by the participant on the scale after intervention at 1-month post baseline
  Participant satisfaction with services will be assessed using the Client Satisfaction. The total score ranges from 8 to 32. Higher scores indicate higher level of satisfaction. Questionnaire (CSQ)

CONTACTS AND LOCATIONS:
Locations (8):
- Pakistan (8):
  - Public schools, Quetta, Balochistan
  - Public schools, Peshawar, KPK
  - Public Schools, Lahore, Punjab Province
  - Public schools, Multan, Punjab Province
  - Public schools, Rawalpindi, Punjab Province
  - Public schools, Hyderābād, Sindh
  - Public schools, Karachi, Sindh
  - Public Schools, Nawabshah, Sindh

IPD SHARING:
Plan to Share IPD: No
Only anonymized data will be shared where necessary such as for the purpose of meta-analysis

REFERENCES:
- [Result] Wasserman C, Hoven CW, Wasserman D, Carli V, Sarchiapone M, Al-Halabi S, Apter A, Balazs J, Bobes J, Cosman D, Farkas L, Feldman D, Fischer G, Graber N, Haring C, Herta DC, Iosue M, Kahn JP, Keeley H, Klug K, McCarthy J, Tubiana-Potiez A, Varnik A, Varnik P, Ziberna J, Postuvan V. Suicide prevention for youth--a mental health awareness program: lessons learned from the Saving and Empowering Young Lives in Europe (SEYLE) intervention study. BMC Public Health. 2012 Sep 12;12:776. doi: 10.1186/1471-2458-12-776. PMID 22971152